CLINICAL TRIAL: NCT05926128
Title: Prospective Study of Treatment Free Remission in Patients With Chronic Myeloid Leukemia in Chronic Phase Who Achieved Deep Molecular Response With Tyrosine Kinase Inhibitors in Real Life Setting in Argentina - (Argentine Stop Trial)
Brief Title: Study of Treatment Free Remission in Patients With Chronic Myeloid Leukemia in Chronic Phase
Acronym: AST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundaleu (Other)
Responsible Party: Principal Investigator, Carolina Pavlovsky, Chief of Clinical Research Area, Fundaleu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Argentina Stop Trial; AST2018 (Other: FUNDALEU)
Record Dates: First submitted 2022-06-02; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: CML
Keywords: DISCONTINUATION

STUDY DESIGN:
Intervention Model Description: multicentre, open-label, uncontrolled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CML patient TKI discontinuation study (Other): Treatment free remission in patients with chronic myeloid leukemia in chronic phase who achieved deep molecular response with tyrosine kinase inhibitors
  Interventions: Drug: Discontinuing treatment with Tyrosine Kinase Inhibitor after enrolment

INTERVENTIONS:
Drug: Discontinuing treatment with Tyrosine Kinase Inhibitor after enrolment — Discontinuing treatment with Tyrosine Kinase Inhibitor after enrolment with a scheduled molecular monitoring until month 24.

SUMMARY:
The principal aim of this study is to evaluate complete molecular remission in patients with chronic myeloid leukemia (CML) in deep molecular response after stopping tyrosine kinase inhibitor (TKI) treatment. The second aim is to characterize the immunological status of patients with CML at the time of TKI interruption and then at 3 months after the interruption.

DETAILED DESCRIPTION:
ARGENTINA STOP TRIAL is a multicentre, open-label, uncontrolled trial to estimate the persistence of molecular remission in patients with chronic phase Chronic Myeloid Leukemia (CML) in Deep Molecular Response after stopping Tyrosine Kinase Inhibitor (TKI)

Primary Objective:

- To identify the proportion of patients who continue on Major Molecular Response after discontinuing treatment with TKI.

Secondary objectives:

* To characterize the immunological status of patients with CML at the time of interruption and then at 3 and 12 months after the interruption.

Tertiary objective: To evaluate the pharmacoeconomic impact of interrupting the treatment.

ELIGIBILITY:
Inclusion criteria:

1. Signed Informed consent.
2. Patients with a diagnosis of CML BCR-ABL positive in CP treated with approved TKI (Imatinib, Nilotinib or Dasatinib) in 1st line or in 2nd line due to intolerance to the 1st line or in 2nd line due to the lack of deep MR with 1st line TKI, which never presented criteria for treatment failure.
3. Age ≥ 18 years
4. ≥ 4 years of treatment with imatinib, nilotinib or dasatinib.
5. Achievement of MR 4.5 in a standardized laboratory (BCR-ABL1 IS ≤ 0.0032%).
6. Evidence of MR 4.5 sustained for ≥ 2 years, as documented in at least 4 tests performed at least 3 months apart.
7. Evidence of typical quantifiable BCR-ABL1 transcript (b3a2 [e14a2] and / or b2a2 [e13a2], typical isoforms of p210).

Exclusion criteria:

1. Patients who previously discontinued TKI and demonstrated recurrence of the disease.
2. Patients with failure to any TKI at any time.
3. Patients who presented accelerated phase or CML in blast crisis at any time.
4. Patients with atypical transcript not quantifiable by RT qPCR
5. BCR-ABL mutation detected at any time during the course of the resistant disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Molecular relapse free survival during 24 months | 24 months
  Molecular relapse free survival, defined as the time from the start of TKI interruption until the loss of the MMR.
  RQ PCR (IS) >0.1% BCR ABL will be considered as loss of MMR

SECONDARY OUTCOMES:
Treatment-free survival during 24 months | 24 months
  Treatment-free survival , defined as the time from the start of TKI interruption to the restart of the TKI.

OTHER OUTCOMES:
Overall survival during 24 months | 24 months
  Overall survival, defined from the day of TKI interruption until date of death, date of last contact or loss of follow-up.
Pharmacoeconomic analysis during 24 months | 24 months
  Calculate the total saving of the included patients un US dollars, considering the costs of TKIs, PCRs performing and medical visits,

CONTACTS AND LOCATIONS:
Locations (1):
- FUNDALEU, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No